CLINICAL TRIAL: NCT07009873
Title: Clinical Application on the R&D Purpose of Wearable Ultrasound Sensors:A Single-Center Prospective Study
Brief Title: Clinical Application of Wearable Ultrasound Sensors
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yu-kun Luo, Clinical Professor, Chinese PLA General Hospital
Other Study IDs: S2025-096-01
Record Dates: First submitted 2025-04-27; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-02

CONDITIONS: DVT - Deep Vein Thrombosis; POCUS
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: This study is designed to assess the non-inferiority of a novel ultrasound imaging technique, rather than to evaluate a therapeutic intervention. — This study is designed to assess the non-inferiority of a novel ultrasound imaging technique, rather than to evaluate a therapeutic intervention.

SUMMARY:
This study aims to develop and evaluate a wearable ultrasound imaging sensor for the early diagnosis and real-time monitoring of various diseases, such as cardiovascular conditions and structural abnormalities of superficial organs. With advancements in medical technology, wearable devices have attracted increasing attention for their portability and real-time capabilities.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 yrs and able to consent
* Relevant diagnosis for study arm (heart failure, lower-limb DVT, or ICU monitoring)
* Adequate acoustic window and intact skin at sensor site

Arm-specific:

* Heart-failure arm: Clinically stable HFrEF or HFpEF on standard therapy
* DVT arm: Imaging-confirmed lower-limb DVT, anticoagulated or scheduled for intervention
* ICU arm: ICU/post-op patient requiring continuous bedside ultrasound

Exclusion Criteria:

* Poor acoustic window preventing interpretable images
* Local skin infection, open wound, or implant/hardware blocking sensor
* Inability to cooperate with monitoring

Arm-specific:

* Heart-failure arm: Acute MI or uncontrolled arrhythmia in past 3 months
* DVT arm: Active bleeding or severe coagulopathy
* ICU arm: Unstable multi-organ failure precluding safe monitoring

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participant recruitment will be conducted by licensed physicians during routine clinical follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Image Quality | Day 1 (Baseline): Measured immediately after first wearable sensor placement
  * Signal-to-Noise Ratio (SNR)
  * Unit: decibels (dB)
  * Contrast-to-Noise Ratio (CNR)
  * Unit: decibels (dB)
Image Quality | Day 1 (Baseline): Measured immediately after first wearable sensor placement
  * Axial Resolution
  * Unit: millimeters (mm)
  * Lateral Resolution
  * Unit: millimeters (mm)

SECONDARY OUTCOMES:
Consistency of image quality | Day 1 (Baseline): Measured immediately after first wearable sensor placement
  Image Clarity Score Unit: 5-point Likert scale (1 = poor to 5 = excellent)
Consistency of image quality | Day 1 (Baseline): Measured during the initial imaging session
  Intra-session Reproducibility of SNR Unit: Intraclass correlation coefficient (ICC)
Consistency of image quality | Day 1 (Baseline): Measured during the initial imaging session
  Diagnostic Sensitivity Unit: percent (%)

CONTACTS AND LOCATIONS:
Overall Officials: Yukun Luo, Professor, M.D., Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No